CLINICAL TRIAL: NCT00689702
Title: Cetuximab (Erbitux®), Capecitabine and Radiotherapy in Neoadjuvant Treatment of Patients With Locally Advanced Resectable Rectal Cancer: A Phase II Pilot Study
Brief Title: Cetuximab (Erbitux®), Capecitabine and Radiotherapy in Neoadjuvant Treatment of Patients With Rectal Cancer
Acronym: XERT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Vaneja Velenik, PhD, MD,, Institute of Oncology Ljubljana, Slovenia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-688
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Rectal Cancer
Keywords: cetuximab; capecitabine; radiotherapy; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cetuximab, capecitabine — Cetuximab 400mg/m2 in iv infusion as an initial dose on day 15, then a weekly dose of 250mg/m2 for 5 weeks during radiotherapy (days 22, 29, 36, 43, 50).
  Capecitabine: 1250 mg/m² bd for 14 days (1 cycle); 825mg/m2 bd over 5 weeks during radiotherapy.
  Radiotherapy: planned total dose of 45 Gy in 25 fractions using a four-field plan in 5 weeks.
  Other Names: Erbitux; Xeloda

SUMMARY:
This is a nonrandomised pilot trial to establish the role of intravenous cetuximab when added to a schedule of capecitabine plus pelvic radiation in patients who have locally advanced primary resectable rectal cancers.

DETAILED DESCRIPTION:
Preoperative radiotherapy and 5-FU based chemotherapy, along with the complete resection of the mesorectum is a standard treatment of locally advanced rectal cancer.Capecitabine has the potential to replace 5-FU as standard agent. Cetuximab is a monoclonal antibody directed against EGFR. Both agents are active in treatment of colorectal cancer and have demonstrated radiosensitising properties.The trial aims to assess the efficacy, safety and toxicity of the combination of cetuximab, capecitabine and radiation in patients with stage II and III rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 if judged fit for surgery
* WHO performance status 0-1
* Histologically proven rectal adenocarcinoma located below the peritoneum
* T3-T4 or/and nodal involvement determined by rectal ultrasound or computed tomography (CT) or MRI
* No distant metastases
* Adequate haematological, cardiac, liver and renal function
* Signed informed consent
* Appropriate measures for contraception for men and women, if applicable

Exclusion Criteria:

* Prior radio- and/or chemotherapy
* Others synchronous cancers
* History of other malignant disease
* Significant heart disease
* Known hypersensitivity to biological drugs
* Pregnant or lactating patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Complete pathological remission rate | at pathological examm of surgical speciment

SECONDARY OUTCOMES:
Rate of sphincter sparing surgical procedure Toxicity/safety | Toxicity/safety:during preoperative treatment, early and late postoperative follow up

CONTACTS AND LOCATIONS:
Overall Officials: Vaneja Velenik, PhD, MD, Principal Investigator — Institute of Oncology, Ljubljana, Slovenia
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia, Slovenia

REFERENCES:
- [Background] Kim JC, Kim TW, Kim JH, Yu CS, Kim HC, Chang HM, Ryu MH, Park JH, Ahn SD, Lee SW, Shin SS, Kim JS, Choi EK. Preoperative concurrent radiotherapy with capecitabine before total mesorectal excision in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):346-53. doi: 10.1016/j.ijrobp.2005.02.046. PMID 15913913
- [Background] Grunwald V, Hidalgo M. Development of the epidermal growth factor receptor inhibitor Tarceva (OSI-774). Adv Exp Med Biol. 2003;532:235-46. doi: 10.1007/978-1-4615-0081-0_19. PMID 12908562
- [Background] Velenik V, Anderluh F, Oblak I, Strojan P, Zakotnik B. Capecitabine as a radiosensitizing agent in neoadjuvant treatment of locally advanced resectable rectal cancer: prospective phase II trial. Croat Med J. 2006 Oct;47(5):693-700. PMID 17042060
- [Background] Robert F, Ezekiel MP, Spencer SA, Meredith RF, Bonner JA, Khazaeli MB, Saleh MN, Carey D, LoBuglio AF, Wheeler RH, Cooper MR, Waksal HW. Phase I study of anti--epidermal growth factor receptor antibody cetuximab in combination with radiation therapy in patients with advanced head and neck cancer. J Clin Oncol. 2001 Jul 1;19(13):3234-43. doi: 10.1200/JCO.2001.19.13.3234. PMID 11432891